CLINICAL TRIAL: NCT01389830
Title: End of Life Treatment Preferences of Latino Medicare Beneficiaries With Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2011-0436; 7K01CA151785-02 (NIH)
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Advanced Cancers
Keywords: End of Life; EOL; Latinos; Hispanic American; Medicare beneficiaries; stage III diagnosis; Breast cancer; Colorectal cancer; Prostate cancer; Lung cancer; Cancer Prevention and Treatment Demonstration; CPTD
MeSH Terms: conditions — Death; Disease; Breast Neoplasms; Colorectal Neoplasms; Prostatic Neoplasms; Lung Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Older Latinos With Cancer: Monthly Telephone Survey of Cohort with stage III or greater of breast, colorectal, or prostate cancer up until 12 months.
  Interventions: Behavioral: Telephone Survey
- Older Latinos Without Cancer: Single Telephone Survey of Cohort without a history of cancer.
  Interventions: Behavioral: Telephone Survey

INTERVENTIONS:
Behavioral: Telephone Survey — Telephone interviews (survey) at baseline taking approximately 30-40 minutes to complete; follow-up monthly surveys for cancer patients take 20-30 minutes to complete, follow ups until 12 months or death.
  Other Names: Interviews

SUMMARY:
Objectives:

The primary objective of the research project is to investigate how declining health status influences the end-of-life (EOL) treatment preferences in Latino Medicare beneficiaries with cancer and to examine if and how these preferences are modified by predisposing characteristics (i.e., acculturation, education, medical mistrust, perceived racism) and/or provider-related characteristics (i.e., ethnicity, language used, provision of interpreters, or patient navigators). The specific aims are:

1. To determine if declining functional status influences the end-of-life treatment preferences of older Latino Medicare beneficiaries with cancer.
2. To determine if predisposing characteristics (i.e., acculturation, age, education, medical mistrust, perceived racism) and/or provider-related characteristics (i.e., ethnicity, language used, provision of interpreters, or patient navigators) modify the association between end-of-life treatment preferences and declining health status in older Latino Medicare beneficiaries with cancer.
3. To identify if the end-of-life treatment preferences of Latino Medicare beneficiaries with cancer differ from those of older Medicare beneficiaries without cancer.

DETAILED DESCRIPTION:
Latino Medicare Beneficiary With Cancer:

This study will determine if the combination of declining health, cultural factors (such as language of choice) and meeting the cultural and language needs of Latino cancer patients influence end-of-life treatment choices over time.

If participant decides to take part in this study, participant will complete a questionnaire once a month for 9 months, over the telephone. The questionnaire asks participant about participant's end of life and decision making preferences, as well as questions about participant's health status and other basic questions about participant such as participant's education level, age, and health insurance. The first phone questionnaire, the one participant will answer today, will take about 30 - 40 minutes to complete. The monthly surveys after today will take about 20 - 30 minutes to complete each month. Participant will be considered off of the study in nine months.

Should participant become too ill and are unable to complete the surveys, researchers will ask a proxy to respond on participant's behalf. A proxy in this case, should be someone participant trusts, who knows participant well enough to know how to answer the health questionnaire on participant's behalf. A proxy is usually a spouse, child, other close family member or friend. This person will only have to answer questions about participant. He or she will not answer any questions about him or herself. Researchers will ask participant to provide researchers with the contact information of the person participant selects as participant's "questionnaire proxy" today at the end of this consent form. If participant is able to complete all 9 surveys, researchers will not contact the proxy.

Information from this study will be used only for research purposes. All identifying information such as participant's name and address will be kept private. This information may be kept at MD Anderson and University of Houston (UH) forever. Participant will be assigned a code number so that participant's name will not be used. The research team at MD Anderson and UH will be able to link the code number to participant's name. Researchers will take appropriate steps to keep participant's survey responses confidential. However, there is no guarantee of absolute confidentiality. Participant's information will be protected according to state and federal law. The research team may share study information with certain individuals including the National Institutes of Health and institutional study monitors who verify the accuracy of the information to see that the research is being conducted in a safe and correct manner.

Answering the survey questions over the phone may cause participant to feel tired. The questionnaires may involve topics that are sensitive in nature. Participant may refuse to answer any question that makes participant feel uncomfortable. If participant has concerns after completing the survey, participant is encouraged to contact participant's doctor, the study chair, or MD Anderson's Institutional Review Board.

Latino Medicare Beneficiary Without Cancer:

This study will determine if the combination of declining health, cultural factors (such as language of choice) and meeting the cultural and language needs of Latino cancer patients (provider ethnicity, use of interpreters), influence end-of-life treatment choices over time.

If participant decides to take part in this study, participant will complete a one-time questionnaire today, over the telephone. The questionnaire asks participant about participant's end of life and decision making preferences, as well as questions about participant's health status and other basic questions about participant such as participant's education level, age, and health insurance. This questionnaire will take about 30 - 40 minutes to complete. Participant will be considered off the study after participant completes this one-time questionnaire.

Information from this study will be used only for research purposes. All identifying information such as participant's name and address will be kept private. This information may be kept at MD Anderson and University of Houston (UH) forever. Participant will be assigned a code number so that participant's name will not be used. The research team at MD Anderson and UH will be able to link the code number to participant's name. Researchers will take appropriate steps to keep participant's survey responses confidential. However, there is no guarantee of absolute confidentiality. Participant's information will be protected according to state and federal law. The research team may share study information with certain individuals including the National Institutes of Health and institutional study monitors who verify the accuracy of the information to see that the research is being conducted in a safe and correct manner.

Answering the survey questions over the phone may cause participant to feel tired. The questionnaires may involve topics that are sensitive in nature. Participant may refuse to answer any question that makes participant feel uncomfortable. If participant has concerns after completing the questionnaires and interviews, participant is encouraged to contact participant's doctor or the study chair.

ELIGIBILITY:
Inclusion Criteria:

1. (Inclusion Criteria of participants recruited from CPTD) Cancer and non-cancer participants recruited to the study must have either been enrolled in either the screening (cancer negative) or treatment (cancer positive) of the Centers for Medicare and Medicaid Services Cancer Prevention and Treatment Demonstration Project (CMS CPTD) (Protocol 2006-0419) or must be listed as a current patient from the provided MD Anderson Tumor Registry list. All participants must meet the CPTD eligibility criteria listed below.
2. (Inclusion Criteria of participants recruited from CPTD) Cancer patients must have a stage III diagnosis or greater of cancer.
3. (Inclusion Criteria of participants recruited from the CPTD) Cancer patients must designate a proxy respondent at the time of the baseline interview in the event that a participant cannot complete subsequent phone interviews due to illness severity or cognitive impairment.
4. (Inclusion Criteria of the CPTD, Protocol 2006-0419) All participants must: Be Latino / Hispanic American.
5. (Inclusion Criteria of the CPTD, Protocol 2006-0419) All participants must: Have Medicare Part A and Part B.
6. (Inclusion Criteria of the CPTD, Protocol 2006-0419) All participants must: Be at least 40 years of age.
7. (Inclusion Criteria of the CPTD, Protocol 2006-0419) All Cancer Screening Group (cancer negative) participants must: Be a Medicare-eligible beneficiary from Region 6 (Central Gulf Coast) as defined by Texas Department of State Health Services.
8. (Inclusion Criteria of the CPTD, Protocol 2006-0419) All Cancer Treatment Group (cancer positive) participants must: Have been diagnosed with breast, cervix, prostate, colorectal, and/or lung cancer within the past 5 years. Be a Medicare-eligible beneficiary from Texas.
9. (Inclusion Criteria of participants recruited from Tumor Registry) Be Latino / Hispanic American.
10. (Inclusion Criteria of participants recruited from Tumor Registry) Have Medicare Part A and Part B.
11. (Inclusion Criteria of participants recruited from Tumor Registry) Be at least 40 years of age.
12. (Inclusion Criteria of participants recruited from Tumor Registry) Must have a stage 3 diagnosis of cancer or greater.
13. (Inclusion Criteria of participants recruited from Tumor Registry) Must designate a proxy respondent at the time of the baseline interview in the event that a participant cannot complete subsequent phone interviews due to illness severity or cognitive impairment.

Exclusion Criteria:

1. Participants refuse to participate in the study or are not competent to give informed consent.
2. Participants who miss 3 or more answers on the Six-Item Screener to Identify Cognitive Impairment.
3. Participants are not able to complete the baseline assessment forms.
4. (Exclusion Criteria of the CPTD, Protocol 2006-0419) All participants must: Not be enrolled in a managed care plan (also called an HMO, Medicare + Choice, or Medicare Advantage)
5. (Exclusion Criteria of the CPTD, Protocol 2006-0419) All participants must: Not be enrolled in hospice
6. (Exclusion Criteria of the CPTD, Protocol 2006-0419): All Cancer Screening Group (cancer negative) participants must: Not have been diagnosed with cancer within the last 5 years.
7. (Exclusion Criteria of the CPTD, Protocol 2006-0419): All Cancer Treatment Group (cancer positive) participants must: Not Be a Medicare-eligible beneficiary outside of Region 6 (Central Gulf Coast) unless treated at MD Anderson.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Survey of 200 older Latino Medicare beneficiaries from the greater Houston area enrolled in a larger national Cancer Prevention and Treatment Demonstration Project (CPTD).
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2011-06-30 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
End of Life Treatment Preferences of Older Latinos With and Without Cancer (Survey Responses) | Once a month for 12 months
  Survey of how changes in functional status influence End of Life (EOL) treatment preferences among older Latinos with cancer. EOL treatment preferences treated as a continuous variable (0-10) and functional status assessed using Patient-reported Eastern Cooperative Oncology Group (ECOG) Performance Scale where low functional status will be defined as an ECOG score of 3 or 4 and high as 0-2.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Torres, MPH, DRPH, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org